CLINICAL TRIAL: NCT01941459
Title: Comparison of Blood Cardioplegia and Custodiol on Patients Operated for Significant Mitral Valve Innsufisiens. An Prospective, Randomized Two-center Study.
Brief Title: Comparison of Blood Cardioplegia and Custodiol
Status: Completed | Type: Observational
Sponsor: Ullevaal University Hospital (Other)
Responsible Party: Principal Investigator, Bjørn Braathen, MD. Ph.D, Oslo University Hospital
Organization: Oslo University Hospital (Other)
Other Study IDs: 2007-001780-30
Record Dates: First submitted 2012-05-07; First posted 2013-09-13 (Estimated); Last update posted 2013-09-13 (Estimated); Status verified 2013-09

CONDITIONS: Mitral Insufficiencies; Myocardial Protection
Keywords: CK-MB; troponin-T

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 1 Custodiol: Custodiol
- 2 Blood cardioplegia: Blood cardioplegia

SUMMARY:
Thru the last 20 years it has been a discussion witch solution that gives the best myocardial protection during cardiac arrest by heart operations.

* It has been a tendency that a blood based cardioplegia gives a better protection bye long ischemic times but it has not been possible too conclude in this matter.
* The investigators have two groups of cardioplegia, the blood based and, the crystalloid based cardioplegia.
* It has been done a lot of studies to see what kind of cardioplegia that gives the best myocardial protection. Different temperature, different amount and content, retrograde or antegrade or both, contentiously and further on have been tested without a clear conclusion.
* The investigators decided to make a study with a cohort of patients as homogenous as possible with a cross clamp time around 70 min.
* Adult patients' with a severe aortic stenoses without any other significant heart disease was included in our prospective randomised study.
* Patients with additional significant coronary artery disease (≥ 50% stenoses) were excluded from the study.
* The investigators used the well known biomarkers CK-MB and troponin-T too evaluate the myocardial damage.

DETAILED DESCRIPTION:
Objective: Myocardial protection during a cardiac arrest is mostly managed with cardioplegia. To day we normally used a blood or crystalloid based solutions. It has been published a lot of papers comparing the too groups with different results. To our knowledge no prospective, randomized study has compared modified St Thomas based Blood and Crystalloid cardioplegia on the acknowledged markers (CK-MB, troponin-T) of myocardial damage during aortic valve replacement on patients without additional significant coronary artery disease.

Methods: 100 patients with aorta stenoses undergoing aortic valve replacement without significant coronary artery stenoses or other significant concomitant heart valve disease were included in the study. They were given antegrade cold blood or cold crystalloid cardioplegia delivered through the coronary Ostia every 20 min throughout the period of aortic cross-clamp. CK-MB and troponin-T were compared between the two groups.

Published 2010 in the journal of thoracic and cardiovascular surgery.

ELIGIBILITY:
The study protocol was approved by the local ethical committees. Eligible for operation were:

Inclution Criteria

* patients with mitral regurgitation equal to or larger than grade 3 out of 4.
* Ablation for atrial fibrillation was the only concomitant procedure that was allowed in addition to mitral valve surgery and these patients were block-randomized to ensure equally many patients with ablation in the two groups of cardioplegia.

Exclusion Criteria

* Patients with any other concomitant heart valve disease or coronary artery stenoses (≥ 50%) were excluded from the study.
* Age below 18
* Pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Between Mars 2007 and December 2009, 80 consecutive patients undergoing elective mitral valve surgery for mitral regurgitation at Oslo University Hospital Ullevål, Oslo, Norway and Sahlgrenska University Hospital, Gothenburg, Sweden were included in the study after informed written consent.
Sampling Method: Non-Probability Sample
Enrollment: 76 (Actual)
Dates: Start 2007-03; Primary Completion 2009-12 (Actual); Study Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
CK-MB ,troponin-T | 72 hours

CONTACTS AND LOCATIONS:
Overall Officials: Theis Tønnessen, prof.dr.med, Study Director — Thoraxkirurgisk avd. UUS; Bjørn Braathen, med.doc, Study Chair — Thoraxkir.avd. UUS
Locations (1):
- thoraxkirurgisk avd, UUS, Oslo, Norway